CLINICAL TRIAL: NCT05097365
Title: Effect of Methyl-donor Nutrient Supplementation on Methylation Profile of Inflammatory-related Genes in Lupus Patients With Obesity: a Clinical Trial
Brief Title: Methyl-donor Nutrient Supplementation and Methylation Profile in Lupus Patients With Obesity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SLE and DNA methylation
Record Dates: First submitted 2021-08-10; First posted 2021-10-28 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity; Lupus Erythematosus
MeSH Terms: conditions — Overweight; Obesity | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Supplemented Normal Weight Group (Experimental): Patients with normal weight (BMI between 18.5 and 24.9 kg/m²) that will receive supplementation.
  Interventions: Dietary Supplement: Vitamin B12 + folic acid supplementation
- Supplemented Excess Body Weight Group (Experimental): Patients with excess body weight (BMI > 25 kg/m²) that will receive supplementation.
  Interventions: Dietary Supplement: Vitamin B12 + folic acid supplementation
- Control Normal Weight Group (Placebo Comparator): Patients with normal weight (BMI between 18.5 and 24.9 kg/m²) that will receive placebo.
  Interventions: Dietary Supplement: Placebo supplementation
- Control Excess Body Weight Group (Placebo Comparator): Patients with excess body weight (BMI > 25 kg/m²) that will receive placebo.
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin B12 + folic acid supplementation — A 12 weeks parallel-group randomised controlled trial will be performed, in which erythematous lupus patients will complete a vitamin B12 and folic acid supplementation, in addition to the usual therapy. The dietary supplementation will be by capsules, which will content 400 mcg of folic acid and 2000 mcg of vitamin B12 each.
  Arms: Supplemented Excess Body Weight Group; Supplemented Normal Weight Group
Dietary Supplement: Placebo supplementation — A 12 weeks parallel-group randomised controlled trial will be performed, in which erythematous lupus patients will complete a placebo supplementation.The placebo and vitamin B12 + folic acid supplement will be indistinguishable in terms of taste, smell, and appearance.
  Arms: Control Excess Body Weight Group; Control Normal Weight Group

SUMMARY:
Dietary supplementation with methyl donors has been demonstrated to increase DNA methylation in leucocytes whereas a limited dietary intake of methyl donors was associated with DNA hypomethylation. Considering SLE disease, previously study showed that high doses of vitamin B6 and folate were associated with less severe SLE. Furthermore, some evidences reported a relatively high incidence of decreased serum B12 levels in rheumatic patients. This led to the suggestion that diets rich in methyl group donors could have beneficial effects on SLE.

ELIGIBILITY:
Inclusion criteria:

* SLE diagnosis
* Female
* In pre-menopausal period
* Aged between 18 to 45 years
* Patients that meet the classification criteria according to Systemic Lupus International Collaborating Clinics classification criteria (SLICC)
* Patients with SLEDAI score ≤ 4 on Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K)
* Under prednisone treatment at a dosage <10 mg/day
* Under treatment with chloroquine at a stable dose
* BMI > 18,5 kg/m2

Exclusion Criteria:

* Current infection
* Diabetes
* Arterial hypertension
* Smokers
* Pregnancy
* Anticoagulants use
* Methotrexate use
* Other autoimmune diseases
* Current vitamin B12 or/and folic acid supplementation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on DNA methylation profile at 12 weeks | Baseline and 12 weeks
  Percentage of DNA methylation level
Change from baseline on weight at 12 weeks | Baseline and 12 weeks
  Weight in kilograms
Change from baseline on serum vitamin B12 concentrations at 12 weeks | Baseline and 12 weeks
  Serum vitamin B12 concentrations in pg/mL
Change from baseline on serum folic acid concentrations at 12 weeks | Baseline and 12 weeks
  Serum folic acid concentrations in ng/mL

SECONDARY OUTCOMES:
Age of onset | Baseline
  Units of Measure: years
Duration of disease since diagnosis | Baseline
  Units of Measure: years
Change from baseline on miR-146 expression at 12 weeks | Baseline and 12 weeks
  Relative miR-146 expression
Change from baseline on miR-181 expression at 12 weeks | Baseline and 12 weeks
  Relative miR-181 expression
Change from baseline on miR-21 expression at 12 weeks | Baseline and 12 weeks
  Relative miR-21 expression
Change from baseline on miR-126 expression at 12 weeks | Baseline and 12 weeks
  Relative miR-126 expression
Change from baseline on TNF-a gene expression at 12 weeks | Baseline and 12 weeks
  Relative gene expression of TNF-a
Change from baseline on LEP gene expression at 12 weeks | Baseline and 12 weeks
  Relative gene expression of LEP
Change from baseline on ADIPOQ gene expression at 12 weeks | Baseline and 12 weeks
  Relative gene expression of ADIPOQ
Change from baseline on MTHFR gene expression at 12 weeks | Baseline and 12 weeks
  Relative gene expression of MTHFR
Change from baseline on STAT3 gene expression at 12 weeks | Baseline and 12 weeks
  Relative gene expression of STAT3
Change from baseline on IL-6 gene expression at 12 weeks | Baseline and 12 weeks
  Relative gene expression of IL-6
Change from baseline on DNMT1 gene expression at 12 weeks | Baseline and 12 weeks
  Relative gene expression of DNMT1
Change from baseline on serum leptin concentrations at 12 weeks | Baseline and 12 weeks
  Serum leptin concentration in ng/mL
Change from baseline on serum IL-6 concentrations at 12 weeks | Baseline and 12 weeks
  Serum IL-6 concentration in ng/mL
Change from baseline on serum IL-17 concentrations at 12 weeks | Baseline and 12 weeks
  Serum IL-17 concentration in ng/mL
Change from baseline on serum IL-2 concentrations at 12 weeks | Baseline and 12 weeks
  Serum IL-2 concentration in ng/mL
Change from baseline on serum TNF-a concentrations at 12 weeks | Baseline and 12 weeks
  Serum TNF-a concentration in ng/mL
Change from baseline on serum C-reactive protein concentrations at 12 weeks | Baseline and 12 weeks
  Serum C-reactive protein concentration in ng/mL
Change from baseline on serum adipokines concentrations at 12 weeks | Baseline and 12 weeks
  Serum adipokines concentration in ng/mL
Change from baseline on serum triglycerides concentrations at 12 weeks | Baseline and 12 weeks
  Serum triglycerides concentration in mg/dL
Change from baseline on serum cholesterol concentrations at 12 weeks | Baseline and 12 weeks
  Serum cholesterol concentrations in mg/dL
Change from baseline on serum glucose concentrations at 12 weeks | Baseline and 12 weeks
  Serum glucose concentrations in mg/dL
Change from baseline on dietary intake at 12 weeks | Baseline and 12 weeks
  Dietary intake in g and percentage
Change from baseline on abdominal circumference at 12 weeks | Baseline and 12 weeks
  Abdominal circumference in centimeters
Change from baseline on fat mass at 12 weeks | Baseline and 12 weeks
  Fat mass in kilograms
Change from baseline on fat free mass at 12 weeks | Baseline and 12 weeks
  Fat free mass in kilograms
Change from baseline on body mass index at 12 weeks | Baseline and 12 weeks
  Body mass index in kilograms/meters^2
Change from baseline on height at 12 weeks | Baseline and 12 weeks
  Height in meters

CONTACTS AND LOCATIONS:
Locations (1):
- Univsersity of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Carvalho LM, da Mota JCNL, Ribeiro AA, Souza LL, Sposeto RB, Pinhel MAS, Nonino CB, Costa-Fraga N, Crujeiras AB, Izquierdo AG, Diaz-Lagares A, Hounkpe BW, Borba EF, Gualano B, Nicoletti CF. Epigenetic and metabolic signatures in systemic lupus erythematous: The impact of excess body weight on adipose tissue DNA methylation profile. Genomics. 2026 Feb 8;118(2):111217. doi: 10.1016/j.ygeno.2026.111217. Online ahead of print. PMID 41666998
- [Derived] da Mota JCNL, Carvalho LM, Souza LL, Ribeiro AA, Pinhel MAS, Nonino CB, Godoy AL, Borba EF, Hounkpe BW, Gualano B, Nicoletti CF. Nutritional status-dependent DNA methylation modifications on adipose tissue in systemic lupus erythematosus women following folic acid and vitamin B12 supplementation: a randomized double-blind placebo-controlled trial. Clin Epigenetics. 2026 Jan 3. doi: 10.1186/s13148-025-02041-5. Online ahead of print. PMID 41484640
- [Derived] da Mota JCNL, Carvalho LM, Ribeiro AA, Souza LL, Borba EF, Roschel H, Gualano B, Nicoletti CF. Methyl-donor supplementation in women with systemic lupus erythematosus with different nutritional status: the protocol for a randomised, double-blind, placebo-controlled trial. Lupus Sci Med. 2024 Oct 7;11(2):e001279. doi: 10.1136/lupus-2024-001279. PMID 39375179